CLINICAL TRIAL: NCT04465851
Title: The Effect of HydroCurc™ Curcumin and Ferrous Iron Supplementation on Iron Status and Inflammatory and Neurotrophic Marker Levels in Healthy Adults
Brief Title: Effect of Ferrous iROn and cUrcumin sTatus on Inflammatory and Neurotrophic markErs
Acronym: Fe-ROUTINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: Gencor Pacific Group (Industry)
Responsible Party: Principal Investigator, Mohammed Gulrez Zariwala, Reader in Translational Physiology, University of Westminster
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: ETH1718-0907
Record Dates: First submitted 2020-06-23; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: nutraceutical; anti-oxidant; oxidative status; ferrous sulphate; curcumin; inflammatory status; turmeric; gastrointestinal; fatigue; iron; Hydrocurc; supplement
MeSH Terms: conditions — Iron Deficiencies; Fatigue | interventions — ferrous sulfate; Curcumin; turmeric extract

STUDY DESIGN:
Intervention Model Description: Allocation: Randomisation (block) Intervention Model: Parallel, Randomised placebo-controlled design Masking: Double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants (and supplements) will be coded and randomly allocated (applied randomly by software [gender balanced[) to treatment arms to eliminate order effects and maintain research staff blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- FS65_Curc (Active Comparator): Ferrous Sulphate (65 mg/day elemental iron) and Curcumin 500 mg/day
  Interventions: Dietary Supplement: Ferrous Sulphate 65 mg; Dietary Supplement: Curcumin
- FS65_Plac (Placebo Comparator): Ferrous Sulphate (65 mg/day elemental iron) and Placebo (Curcumin placebo [cellulose])
  Interventions: Dietary Supplement: Ferrous Sulphate 65 mg; Other: Placebo (Curcumin)
- FS0_Plac (Placebo Comparator): Placebo (Ferrous Sulphate placebo [cellulose]) and Placebo (Curcumin placebo [cellulose])
  Interventions: Other: Placebo (Ferrous Sulphate); Other: Placebo (Curcumin)
- FS18_Plac (Placebo Comparator): Ferrous Sulphate (18 mg/day elemental iron) and Placebo (Curcumin placebo [cellulose])
  Interventions: Other: Placebo (Curcumin); Dietary Supplement: Ferrous Sulphate 18mg
- FS18_Curc (Active Comparator): Ferrous Sulphate (18 mg/day elemental iron) and Curcumin 500 mg/day
  Interventions: Dietary Supplement: Curcumin; Dietary Supplement: Ferrous Sulphate 18mg

INTERVENTIONS:
Dietary Supplement: Ferrous Sulphate 65 mg — Oral ferrous salt supplement Ferrous Sulphate 200 mg (equiv. 65 mg elemental iron content)
  Participants instructed to swallow opaque capsules with water away from meals (on an empty stomach)
  At the mid-point visit day (day 21) and the finally at the end-point (day 42) compliance will be verified by counting capsules
  Other Names: Ferrous Sulfate
  Arms: FS65_Curc; FS65_Plac
Dietary Supplement: Curcumin — HydroCurc™ 500 mg formulated curcumin
  At the mid-point visit day (day 21) and the finally at the end-point (day 42) compliance will be verified by counting capsules
  Participants instructed to swallow opaque capsules with water away from meals (on an empty stomach)
  Other Names: Turmeric; Curcuma longa
  Arms: FS18_Curc; FS65_Curc
Other: Placebo (Ferrous Sulphate) — Microcrystalline cellulose
  Participants instructed to swallow opaque capsules with water away from meals (on an empty stomach)
  Arms: FS0_Plac
Other: Placebo (Curcumin) — Microcrystalline cellulose
  Participants instructed to swallow opaque capsules with water away from meals (on an empty stomach)
  Arms: FS0_Plac; FS18_Plac; FS65_Plac
Dietary Supplement: Ferrous Sulphate 18mg — Oral ferrous salt supplement
  Ferrous Sulphate 55 mg (equiv. 18 mg elemental iron content)
  Participants instructed to swallow opaque capsules with water away from meals (on an empty stomach)
  At the mid-point visit day (day 21) and the finally at the end-point (day 42) compliance will be verified by counting capsules
  Other Names: Ferrous Sulfate
  Arms: FS18_Curc; FS18_Plac

SUMMARY:
INTRODUCTION: Iron is a vital nutrient for many physiological processes including DNA production, oxygen transport and neuronal processes. However, several factors limit iron absorption including: limited bioavailability of iron (dietary or supplementation sources), can be subject to dietary iron inhibitors (e.g. calcium). Excess iron can cause cellular oxidative stress in the body.

Curcumin is an active component found in turmeric, known for its anti-oxidant and anti-inflammatory properties. Co-administration of iron and curcumin may influence iron, inflammatory status and/or neurotrophic markers in the body.

DETAILED DESCRIPTION:
Intervention study with five parallel treatment groups in a randomised, double-blind, placebo-controlled design.

Study population: Healthy Participants (Male or Female) will receive daily supplements (active or equivalent placebos) for 6 weeks (42 days)

Biological samples (blood and urine samples) are collected at baseline visit (day 1), mid-point (day 21) and end-point (day 42). In addition, pertinent questionnaires (Visual Analogue Scale-Fatigue [VAS-F] and oral iron supplement questionnaire will be collected at the aforementioned time points.

ELIGIBILITY:
Inclusion Criteria:

* Males & Females (18-40 years of age)
* Healthy subjects

Exclusion Criteria:

* <18 years or >40 years
* Dieters
* Consumption of >21 serving of alcohol/week
* Any allergies/health issues related to items being ingested
* Any serious illnesses or those on medication
* Any pregnant or lactating women
* Any women who are trying to conceive
* Any women taking contraceptive medication
* Any gastrointestinal disorders
* Any chronic menstrual disorders
* Any subjects who have undergone the menopause or undergoing the perimenopause transition
* Any eating disorders
* Any depression/mental disorders
* Any abnormal blood pressure levels
* Those with deficient/excess/abnormal iron levels according to United Kingdom (UK) guidelines &/or haemochromatosis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male or Female
Enrollment: 155 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated inflammation | Change in Interleukin 6, Interleukin 10 and Interleukin 1 beta (ELISA) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: Interleukin 6 (pg/mL), Interleukin 10 (pg/mL), Interleukin 1 beta (pg/mL)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated inflammation | Change in Tumour Necrosis Factor alpha (ELISA) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Tumour Necrosis Factor alpha (pg/mL)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated inflammation | Change in C-Reactive Protein (immunoassay) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: C-Reactive Protein (g/L)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated lipid peroxidation | Change in thiobarbituric acid reactive substances (ELISA) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: thiobarbituric acid reactive substances (μM)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated acute iron absorption | Change in serum iron (colorimetric analyser) from 0 and 180 minutes following supplementation
  Marker: serum iron (μmol/L)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated acute iron absorption | Change in total iron binding capacity (colorimetric analyser) from 0 and 180 minutes following supplementation
  Marker: total iron binding capacity (μmol/L)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated iron status | Change in serum iron (colorimetric analyser) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: serum iron (μmol/L)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated iron status | Change in total iron binding capacity (colorimetric analyser) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: total iron binding capacity (μmol/L)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated iron status | Change in ferritin (immunoassay) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: Ferritin (ng/mL)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated iron status | Change in haemoglobin (whole blood analyser) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: Haemoglobin (g/dL)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated iron status | Change in red blood cells (whole blood analyser) from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: Red blood cells (M/μL)

SECONDARY OUTCOMES:
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated neurotrophic levels | Change in BDNF (ELISA) from baseline to endpoint from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Marker: Brain derived neurotrophic factor (BDNF) (ng/mL)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated gastrointestinal effects | Change in reported subjective gastrointestinal effects from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Subjective analysis including: Oral Iron Supplement Questionnaire
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated perception of fatigue | Change in VAS-F from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Subjective analysis including: Visual Analogue Scale for Fatigue (VAS-F). Scores range from 0 to 100 (the higher the score the greater the level of fatigue)
To assess the influence of HydroCurc™ administration on ferrous iron supplementation associated perception of fatigue | Change in FSS from day 1 compared to day 21 (baseline to midpoint), day 1 compared to day 42 (baseline to endpoint) and day 21 compared to day 42 (midpoint to endpoint)
  Subjective analysis including: Fatigue Severity Scale (FSS). The total score of all answers indicates level of fatigue (a total score above ≥ 36 indicates fatigue).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Westminster, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No